CLINICAL TRIAL: NCT06907381
Title: Blood Flow-restricted Resistance Exercise to Promote Muscle Strength and Use in Adults With Incomplete Spinal Cord Injury
Status: Enrolling by invitation | Type: Observational
Sponsor: Quality Living, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: QualityLiving
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injury Cervical
Keywords: Blood flow-restricted resistance exercise; Physical therapy; Rehabilitation; Electrical stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Blood flow-restricted resistance exercise — Participants will engage in baseline measurement of blood pressure, strength of target muscle contractions, and level of support needed for functional task performance. They will then begin BFRE treatment supplemented by electrical stimulation, if needed, two times weekly. Each exercise session will include performance of four sets of 20 repetitions of target muscle contraction on each side of the body followed by functional task performance.
  Other Names: BFRE

SUMMARY:
Recovery of arm and hand motor control is critical for independence and quality of life following incomplete spinal cord injury (iSCI). Blood flow-restricted resistance exercise (BFRE) has emerged as a potential treatment addressing this need, but treatment guidelines and research reporting effectiveness are sparse. The purpose of this work is to provide case reports of people with cervical iSCI who use BFRE supplemented by electrical stimulation (ES) to increase the strength and functional use of selected upper extremity muscles.

ELIGIBILITY:
Inclusion Criteria:

* Incomplete cervical spinal cord injury
* Resting blood pressure between 80/50 mmHg and 150/90 mmHg for at least three consecutive days
* Native speaker of English

Exclusion Criteria:

* Recent history of deep vein thrombosis or cardiovascular disease including uncontrolled hypertension or a blood-clotting disorder
* Routine experience of orthostatic hypotension as defined as a drop in systolic/diastolic blood pressure greater than 20/10 mmHg when engaging in physical activity
* Severe cognitive, communication, or behavioral disorder as determined by treatment team

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will include adults with incomplete cervical spinal cord injury. They will be medically stable and enrolled in Quality Living's rehabilitation program in Omaha, NE, at the time of participation. Level of injury can vary from C3 to C8. Participants will demonstrate sensory and motor function consistent with AIS B, C, or D classification.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in muscle strength | Baseline and end of treatment at a maximum of 6 months
  Change in strength of target muscle(s) contraction as measured in pounds of force using a dynamometer.

SECONDARY OUTCOMES:
Change in number of repetitions of unassisted target muscle(s) contractions | Baseline and end of treatment at a maximum of 6 months
  Tally of the number of target muscle contractions participant can perform during a single treatment session (80 repetitions max) without BFRE or electrical stimulation assistance.
Change in support required to perform functional task | Baseline and end of treatment at a maximum of 6 months
  Professional assessment using the 7-point Functional Independence Measure (1 = total assistance; 7 = complete independence) to rate the level of support a participant requires to perform a functional task.
Change in perceived exertion when performing a functional task | Baseline and end of treatment at a maximum of 6 months
  Participants will use the Borg category-ratio 10 Rating Exertion scale (0 = no exertion; 10 = highest level of effort) to rate the effort they expend to perform a functional task.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Waid, DPT, Principal Investigator — Quality Living, Inc.
Locations (1):
- Quality Living, Inc., Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will only consider sharing data in de-identified form and used in publications or presentations resulting from this research. Given that data will be from case examples, we need to exercise extreme caution to ensure the protection of participant privacy.